CLINICAL TRIAL: NCT05933395
Title: Genetically-informed Therapy for ER+ Breast Cancer in a Post-CDK4/6 Inhibitor Setting: a Phase II Umbrella Study (GERTRUDE)
Brief Title: Genetically-informed Therapy for ER+ Breast Cancer Post-CDK4/6 Inhibitor
Acronym: GERTRUDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Mary D Chamberlin, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY02001800; NCI-2024-09317 (Other: National Cancer Institute)
Record Dates: First submitted 2023-05-25; First posted 2023-07-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: locally recurrent; metastatic; ER+; ER+/HER2-
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Fulvestrant; neratinib; Alpelisib; Everolimus; abemaciclib

STUDY DESIGN:
Intervention Model Description: This study has a non-randomized umbrella design. Participants will be assigned to a treatment arm based on tumor/plasma genetic profiling and treatment history using the primary treatment phase algorithm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A- neratinib and fulvestrant (Experimental): Participants with a qualifying ERBB2 (HER2) mutation will be assigned to Treatment Arm A and given the combination of neratinib and fulvestrant until the end of the primary treatment phase.
  Fulvestrant (500 mg) will be administered by intramuscular injection into the buttocks on Cycle 1 Day 1 and Day 15, and on Day 1 of subsequent Cycles.
  Neratinib will initially be administered orally in 3 tablets (total dose of 120 mg) taken 1 time per day with food on Cycle 1 Days 1-7, in combination with fulvestrant starting on Cycle 1 Day 1 as described above. The dose of neratinib will be increased to 4 tablets (total dose of 160 mg) taken 1 time per day with food on Cycle 1 Days 8-14, and then increased further to 6 tablets (240 mg) taken once daily with food thereafter.
  Interventions: Drug: Fulvestrant; Drug: Neratinib
- Arm B- alpelisib and fulvestrant (Experimental): If a participant does not have a qualifying ERBB2 (HER2) mutation, but they have a qualifying PIK3CA mutation, the subject will be assigned to Treatment Arm B and given the combination of alpelisib and fulvestrant until the end of the primary treatment phase.
  Fulvestrant (500 mg) will be administered by intramuscular injection into the buttocks on Cycle 1 Day 1 and Day 15, and on Day 1 of subsequent Cycles.
  Alpelisib will be administered orally in 2 tablets (total dose of 300 mg) taken 1 time per day with food, in combination with fulvestrant as described above.
  Interventions: Drug: Fulvestrant; Drug: Alpelisib
- Arm C- everolimus and fulvestrant (Experimental): If a subject does not have a qualifying ERBB2 or PIK3CA mutation, but they have a qualifying mutation/alteration in AKT1, MTOR, or PTEN, the subject will be assigned to Treatment Arm C and given the combination of everolimus and fulvestrant until the end of the primary treatment phase.
  Fulvestrant (500 mg) will be administered by intramuscular injection into the buttocks on Cycle 1 Day 1 and Day 15, and on Day 1 of subsequent Cycles.
  Everolimus will be administered orally in 1 tablet (10 mg per tablet) taken 1 time per day, in combination with fulvestrant as described above.
  Interventions: Drug: Fulvestrant; Drug: Everolimus
- Arm D- abemaciclib and fulvestrant (Experimental): If a participant does not have a qualifying mutation/alteration for Arms A/B/C, and the participant does not have mutation or loss of RB1, the subject will be assigned to Treatment Arm D and given the combination of abemaciclib and fulvestrant until the end of the primary treatment phase.
  Fulvestrant (500 mg) will be administered by intramuscular injection into the buttocks on Cycle 1 Day 1 and Day 15, and on Day 1 of subsequent Cycles.
  Abemaciclib will be administered orally in 1 tablet (150 mg) taken 2 times per day, in combination with fulvestrant as described above.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant will be administered intramuscularly into the buttocks in combination with one of the other interventions as outlined above.
Drug: Neratinib — Neratinib will be administered orally in tablet form once daily with food in combination with fulvestrant administration as outlined above.
  Arms: Arm A- neratinib and fulvestrant
Drug: Alpelisib — Alpelisib will be administered orally in tablet form once daily with food in combination with fulvestrant administration as outlined above.
  Arms: Arm B- alpelisib and fulvestrant
Drug: Everolimus — Everolimus will be administered orally in tablet form once daily in combination with fulvestrant administration as outlined above.
  Arms: Arm C- everolimus and fulvestrant
Drug: Abemaciclib — Abemaciclib will be administered orally in tablet form twice daily in combination with fulvestrant administration as outlined above.
  Arms: Arm D- abemaciclib and fulvestrant

SUMMARY:
The purpose of this study is to learn if certain drug combinations are effective treatments for patients with advanced ER+/HER2- who have previously been treated with palbociclib, ribociclib, or abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women ≥18 years of age with metastatic ER+ breast cancer, or with locally recurrent ER+ disease not amenable to therapy for curative intent.
2. Patient must be post-menopausal per NCCN guidelines.
3. Patient must have been treated with a CDK4/6i (either palbobclib, ribociclib, or abemaciclib) alone or in combination with an endocrine agent in the advanced disease setting.

   * Up to 3 lines of therapy following CDK4/6i are permissible.
   * Any number of prior lines of endocrine-containing therapy is permissible.
   * Up to 1 prior line of chemotherapy is permissible.
4. Histologic documentation of ER+ breast cancer by core needle biopsy, fine needle aspiration, incisional biopsy, or surgical biopsy of ≥1 site(s) of metastatic or locally recurrent disease performed as standard of care.

   * Exceptions: patients with bone-dominant metastatic disease, or non-bone metastatic disease in whom a safe and accurate biopsy of recurrent/metastatic disease cannot be readily obtained, with a history of ER+ breast cancer are eligible, and biopsy is not required, providing their primary cancer is consistent with the ER criteria described below.
5. ER+ status defined as ER staining by immunohistochemistry in ≥1% of malignant cell nuclei.
6. Tumor must be HER2-non-amplified as defined by an immunohistochemistry score of 0-1+, or with a FISH ratio <2 if IHC is 2+ or if IHC has not been done (as per ASCO/CAP definitions). In cases of borderline or equivocal HER2 status, eligibility will be determined by the PI.
7. Genetic profiling of a tumor or plasma specimen acquired after disease progression on a CDK4/6i must have been performed in a CAP-accredited, CLIA-certified laboratory using clinically validated methods. Profiling must minimally include analysis of study-relevant alterations in ERBB2, PIK3CA, AKT1, MTOR, PTEN, and RB1.

   * If not done: Profiling of a tumor (preferable) or plasma specimen will be performed as part of the study in the DHMC Pathology Laboratory. A plasma specimen may be obtained for study-specific genetic profiling to direct treatment assignment. Tumor specimens must be obtained outside of this study (e.g., by biopsy).
8. If available, archived tumor tissue must be accessible for research purposes, sufficient to make ≥10 five-micron sections; more tumor tissue is preferred.
9. Radiographic staging performed as standard of care, including specifically either PET/CT, or contrast CT (CAP) and bone scan.
10. Patient must be capable and willing to provide informed written consent for study participation.

Exclusion Criteria:

1. Treatment with abemaciclib in the most recent or current line of therapy.
2. During the study Treatment Phases, no concurrent anti-cancer therapies are allowed with the following exception: anti-resorptive bone therapies (e.g., bisphosphonates, denosumab) are permitted.
3. Any investigational cancer therapy in the last 3 weeks.
4. Known untreated CNS disease, unless clinically stable for ≥ 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical benefit within each arm in patients previously treated with a CDK4/6 inhibitor. | 6 - 12 months
  Clinical benefit rate will be measured as the proportion of participants who experience stable disease (SD) at 24 weeks, complete response, and partial response per RECIST 1.1.

SECONDARY OUTCOMES:
Incidence rate of adverse events within each treatment arm. | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE within each treatment arm.
Progression-free survival within each treatment arm. | 12 months
  Progression-free survival will be measured by the time between the initiation of study treatment to the time of progression per RECIST 1.1.
Rate of objective response within each treatment arm. | 12 months
  The proportion of participants within each arm who experience objective response defined as complete or partial response per RECIST 1.1 while on study treatment will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No